CLINICAL TRIAL: NCT06287255
Title: Feasibility and Acceptability of Incorporating Fitbit Smartwatches Into a Health System Referral Based Exercise is Medicine Program in Older Individuals (EIM+)
Brief Title: Feasibility and Acceptability of Incorporating Smartwatches Into an Exercise is Medicine Program in Older Individuals
Acronym: EIM+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Associate Professor of Internal Medicine, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023H0314
Record Dates: First submitted 2024-02-05; First posted 2024-03-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Physical Inactivity; Obesity
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: A single-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise is Medicine Plus (Experimental): Participants receiving the Exercise is Medicine program along with a smartwatch.
  Interventions: Behavioral: EIM+

INTERVENTIONS:
Behavioral: EIM+ — The Exercise is Medicine (EIM) program involves a personalized exercise prescription and wellness coaching component. At the first 1:1 session, participants are provided with a Fitbit and onboarded with Fitabase, allowing for documentation of baseline health behaviors. Over the course of the program, the EIM fitness specialist reviews Fitbit data and progress towards goals, sending push notifications for encouragement and reminders. A personal training session is conducted, followed by sixteen group sessions including up to eight participants. The final session includes updating goals, incorporating Fitbits, and providing an updated exercise prescription. Upon program completion, participants will attend monthly webinars and health coaching sessions at 6- and 12-months post-program. The program aims to help individuals overcome barriers and maintain long-term exercise self-efficacy.

SUMMARY:
The effects of exercise on prevention and improved control of chronic diseases, reduced mortality, and improved quality of life are well established. Exercise has been shown to prevent heart disease, stroke, type 2 diabetes, depression, and certain types of cancers. In addition to prevention, physical activity is included in the standard or care for many chronic diseases and used in treatment. For example, the American Diabetes Association has identified positive health behaviors like physical activity as foundational in the treatment and management of disease and improving overall quality of life.

The Ohio State University Wexner Medical Center Exercise is Medicine Program (EIM) is a physician referral program that aims to increase physical activity to prevent and reduce complications from chronic disease.

The integration of technology among a 65+ population of EIM participants provides a novel approach to improving individual's health. Thus, our study aims to provide EIM participants aged 65+ with smartwatches in the hopes of increasing their overall physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* No healthcare provider-imposed limitations on physical activity
* English-speaking

Exclusion Criteria:

* Symptoms suggestive of coronary artery disease (CAD) or congestive heart failure (CHF) (i.e. chest pain, dizziness, syncope, excessive dyspnea on exertion)
* Myocardial infarction within the last 12 months
* Revascularization within the last 12 months
* Stroke/transient ischemic attack (TIA) within the past 12 months
* Unstable angina
* Congestive heart failure (New York Heart Association (NYHA) Class II, III or IV)
* Ventricular arrhythmia
* Clinically significant cardiac valve disease
* Blood pressure >160/100 mmHg
* Uncontrolled seizure disorder
* Major surgery within the past three months
* Severe or frequent hypoglycemia
* Inability to independently manage blood glucose during activity
* Severe autonomic or peripheral neuropathy
* Active foot ulcers
* Unstable retinopathy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of EIM+ | 12 months
  The co-primary outcome is to determine the feasibility of utilizing smartwatches among Exercise is Medicine participants aged 65+ as assessed by the number of eligible referrals agreeing to participate in the intervention, program attendance, and completion rates.
Acceptability of EIM+ | 12 months
  The co-primary outcome is to determine the acceptability of utilizing smartwatches among Exercise is Medicine (EIM) participants aged 65+ as assessed by survey responses on perception of wearable devices integrated in to the EIM program and program attendance and completion rates.

SECONDARY OUTCOMES:
Change in physical activity | 12 months
  The secondary outcome of physical activity levels before, during and after program completion (preliminary efficacy) will be examined both continuously (moderate-vigorous physical activity minutes per week) and categorically (meeting the goal of 150 minutes of moderate-vigorous physical activity per week).
Change in weight | 12 months
  The secondary outcome is weight before, during and after program completion
Change in BMI | 12 months
  The secondary outcome is BMI before, during and after program completion
Change in hip circumference | 12 months
  The secondary outcome is hip circumference before, during and after program completion
Change in waist circumference | 12 months
  The secondary outcome is waist circumference before, during and after program completion
Change in blood pressure | 12 months
  The secondary outcome is blood pressure before, during and after program completion
Change in heart rate variability | 12 months
  The secondary outcome is heart rate variability before, during and after program completion
Change in hemoglobin A1c | 12 months
  The secondary outcome is hemoglobin A1c before, during and after program completion
Change in perceived stress | 12 months
  The secondary outcome is perceived stress before, during and after program completion as assessed by responses to the Perceived Stress Scale assessment.
Change in depressive symptoms | 12 months
  The secondary outcome is depressive symptoms before, during and after program completion as assessed by responses to the Patient Health Questionnaire-9 (PHQ-9)
Change in diet | 12 months
  The secondary outcome is diet before, during and after program completion as assessed by responses to the Mediterranean Eating Pattern for Americans diet adherence screener.
Change in activity minutes per week | 12 months
  The secondary outcome is activity minutes per week before, during and after program completion as assessed by smartwatch tracking.
Change in daily steps total | 12 months
  The secondary outcome is daily steps taken before, during and after program completion as assessed by smartwatch tracking.
Change in measured steps per minute | 12 months
  The secondary outcome is measured steps per minute before, during and after program completion as assessed by smartwatch tracking.
Change in sleep quality | 12 months
  The secondary outcome is sleep quality before, during and after program completion as assessed by smartwatch tracking.
Change in sleep duration | 12 months
  The secondary outcome is sleep duration before, during and after program completion as assessed by smartwatch tracking.
Change in estimated energy expenditure | 12 months
  The secondary outcome is estimated energy expenditure before, during and after program completion as assessed by smartwatch tracking.
Change in heart rate | 12 months
  The secondary outcome is heart rate before, during and after program completion as assessed by smartwatch tracking.
Change in distance moved | 12 months
  The secondary outcome is distance moved before, during and after program completion as assessed by smartwatch tracking.
Change in minutes of vigorous activity | 12 months
  The secondary outcome is minutes of vigorous activity before, during and after program completion as assessed by smartwatch tracking.
Change in minutes of moderate activity | 12 months
  The secondary outcome is minutes of moderate activity before, during and after program completion as assessed by smartwatch tracking.
Change in minutes of light activity | 12 months
  The secondary outcome is minutes of light activity before, during and after program completion as assessed by smartwatch tracking.
Change in minutes of sedentary time | 12 months
  The secondary outcome is minutes of sedentary time before, during and after program completion as assessed by smartwatch tracking.
Change in number of manually entered and automatically detected physical activities (walking, running, etc.) | 12 months
  The secondary outcome is manually entered and automatically detected physical activities (walking, running, etc.) before, during and after program completion as assessed by smartwatch tracking.
Change in quality of life measures | 12 months
  The secondary outcome is quality of life measures before, during and after program completion as assessed by responses to the RAND Short Form (RAND-SF 36) v1.0 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Joseph, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauben J, Luthy J, Nafiu T, Brengartner A, Omar M, Nemati D, Zhao S, Brock G, Urse K, Paro J, Joseph JJ. Rationale for the Feasibility and Acceptability of Smartwatch Technology in an Exercise Regimen (FASTER) study in older individuals. Contemp Clin Trials. 2026 Jan;160:108152. doi: 10.1016/j.cct.2025.108152. Epub 2025 Nov 18. PMID 41265833